CLINICAL TRIAL: NCT03188757
Title: The Influence of Acute Hyperglycaemia on Oxidative Stress, Inflammation, Neurochemical Profile in Brain and Executive Functions of Adolescents With Type 1 Diabetes Mellitus
Brief Title: The Influence of Acute Hyperglycaemia on Brain in T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Principal Investigator, Tadej Battelino, prof. dr. Tadej Battelino, MD, University of Ljubljana, Faculty of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Hyperglycemia-01
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Hyperglycemia; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- hyperglycaemic clamp (Experimental)
  Interventions: Other: hyperglycaemic clamp

INTERVENTIONS:
Other: hyperglycaemic clamp — 2h hyperglyceamic clamp

SUMMARY:
The study is going to include 20 adolescents, 5-10 years after onset of T1D, aged 12-20 years, on insulin pump. The participants are going to have MRI of the head in euglycaemic and hyperglycaemic state. During both MRI, the participants are going to preform Flanker test, Tower of London test and Spatial memory test. The investigators are going to evaluate the response of inflammation markers and oxidative stress marekers in blood during hypreglycaemia.

DETAILED DESCRIPTION:
The study is going to include 20 patientswith T1D. The group of patients is going to be homogeneous. The inclusion criteria are going to be: duration of T1D approximately 5 - 10 years, age between 10 and 24 years, without associated clinical complications of T1D, similar value of HbA1c and BMI within the normal range (depending on the percentile for age and sex), treatment with an insulin pump. Only the patients who are going to give written consent to participate in the form "Declaration of conscious and free consent" are going to be included.

All selected clinical data to determine the phenotypic characteristics of the patient will be obtained from available medical records or. at their regular outpatient reading.

After 12-hour fasting overnight, the patients will undergo 2h hyperglycaemic clamp.

During hyperglycemia a sample of venous blood for the evaluation of oxidative stress, inflammatory response and the expression of non-coding RNA is going to be drawn.

Subjects will have 1H-MRS in hyperglycaemic and euglycaemic state and evaluation of executive function (using psychological tests) is going to be preformed. For 1H-MRS, the MRI of the head in order to obtain anatomical data is going to be preformed at first .

ELIGIBILITY:
Inclusion Criteria:

* T1D on insulin pump, no diabetic complication, normal BMI and blood pressure

Exclusion Criteria:

-

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
prolonged reaction time | during the MRI in hyperglycaemia

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Faculty - University of Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Suput Omladic J, Slana Ozimic A, Vovk A, Suput D, Repovs G, Dovc K, Bratina N, Avbelj Stefanija M, Battelino T. Acute Hyperglycemia and Spatial Working Memory in Adolescents With Type 1 Diabetes. Diabetes Care. 2020 Aug;43(8):1941-1944. doi: 10.2337/dc20-0171. Epub 2020 May 29. PMID 32471909